CLINICAL TRIAL: NCT05046496
Title: Transplant Renal Artery Stenosis: Observation Versus Stenting - a Feasibility Study
Brief Title: Transplant Renal Artery Stenosis: Observation Versus Stenting
Acronym: TRASOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20HH6286
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Transplant Renal Artery Stenosis
Keywords: Kidney transplant; Transplant renal artery stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational arm (No Intervention): Patients recruited to this arm will undergo no intervention.
- Interventional arm (Active Comparator): Patients recruited to this arm will undergo intra-arterial digital subtraction angiography, with or without intra-arterial stent placement
  Interventions: Diagnostic Test: Intra-arterial digital subtraction angiography

INTERVENTIONS:
Diagnostic Test: Intra-arterial digital subtraction angiography — Invasive intra-arterial angiography, with intra-arterial stent placement if a stenosis is confirmed
  Arms: Interventional arm

SUMMARY:
Transplant renal artery stenosis (TRAS) is abnormal narrowing of the main blood vessel to the kidney transplant and has historically been considered a surgical complication. In heart transplantation, it has long been recognised that rejection can cause narrowing of the heart's blood vessels, and that this complication is the leading cause of heart transplant failure. It is reasonable to assume that this process may also occur in kidney transplantation, which could contribute to premature transplant failure. However, in kidney transplantation it is also likely that other factors, such as surgical factors, traditional cardiovascular risk factors and immunological factors, contribute to the development of TRAS. Given that the disease processes that cause TRAS are not fully understood, at present there is no consensus among kidney doctors on the best means of treating patients diagnosed with TRAS. The aim of the proposed study is to investigate the involvement of these different processes in the development of TRAS, and investigate the optimal way to diagnose and manage TRAS.

At present, there is no standard recommendation for how to treat patients with TRAS. This is partly due to the fact that patients with TRAS may have a broad array of symptoms: Some may have no symptoms, other may have problems with high blood pressure or fluid accumulation, and others may have severe transplant dysfunction. In most transplant centres, patient TRAS and severe symptoms will undergo IADSA and a stent will be placed to open the narrowing. However, it is not clear how best to manage patients with TRAS who have mild to moderate symptoms. We propose to recruit 36 such patients to a clinical study and split them into two groups: One group to undergo IADSA with possible stent placement, and one group to be closely observed. We will then compare transplant function, and other outcomes, after one year between the two groups.

DETAILED DESCRIPTION:
Transplant renal artery stenosis (TRAS) is abnormal narrowing of the main blood vessel to the kidney transplant and has historically been considered a surgical complication. In heart transplantation, it has long been recognised that rejection can cause narrowing of the heart's blood vessels, and that this complication is the leading cause of heart transplant failure. It is reasonable to assume that this process may also occur in kidney transplantation, which could contribute to premature transplant failure. However, in kidney transplantation it is also likely that other factors, such as surgical factors, traditional cardiovascular risk factors and immunological factors, contribute to the development of TRAS. Given that the disease processes that cause TRAS are not fully understood, at present there is no consensus among kidney doctors on the best means of treating patients diagnosed with TRAS. The aim of the proposed study is to investigate the involvement of these different processes in the development of TRAS, and investigate the optimal way to diagnose and manage TRAS.

At present, there is no standard recommendation for how to treat patients with TRAS. This is partly due to the fact that patients with TRAS may have a broad array of symptoms: Some may have no symptoms, other may have problems with high blood pressure or fluid accumulation, and others may have severe transplant dysfunction. In most transplant centres, patient TRAS and severe symptoms will undergo IADSA and a stent will be placed to open the narrowing. However, it is not clear how best to manage patients with TRAS who have mild to moderate symptoms. We propose to recruit 36 such patients to a clinical study and split them into two groups: One group to undergo IADSA with possible stent placement, and one group to be closely observed. We will then compare transplant function, and other outcomes, after one year between the two groups.

ELIGIBILITY:
Inclusion Criteria:

- 1. Renal transplant recipient with a diagnosis of TRAS by radiological imaging, and an MDT decision to proceed with diagnostic IADSA.

2. Aged 18 years and over 3. Able to give informed consent

Exclusion Criteria:

- 1. Estimated GFR <10mls/min/1.73m2 or dialysis dependence 2. Contraindication to angiography (e.g. allergy to radiological contrast) 3. Patients with clinical features of severe TRAS (eg. resistant hypertension, pulmonary oedema and/or rapidly deteriorating function).

4. Any condition or co-morbidity which in the investigator's opinion would make the patient ineligible for the trial or unlikely to adhere to trial procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-08-28 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in eGFR between both arms | 1 year
  measure of kidney transplant function

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) | at baseline, then 1, 3, 6 and 12-months following diagnosis
  measure of kidney transplant function
Change in mean arterial blood pressure (BP), systolic BP and diastolic BP | at baseline, then 1, 3, 6 and 12-months following diagnosis
  Measure of cardiovascular health
Average number of anti-hypertensive medications | at baseline, then 1, 3, 6 and 12-months following diagnosis
  measure of cardiovascular health
Urinary protein : creatinine ratio (UPCR) measurement | at baseline, then 1, 3, 6 and 12-months following diagnosis
  measure of proteinuria
Donor-specific antibody (DSA) free survival | 1 year
  measure of time free from presence of donor-specific antibody in participant's serum
Rejection free survival | 1 year
  measure of time free from histologically proven kidney transplant rejection
Renal allograft failure | 1 year
  Measure of time free from kidney transplant failure
Patient survival | 1 year
  measure of patient survival
Requirement for intervention (primary angiogram in observational group, secondary angiogram in interventional group) | 1 year
  Quantification of patients that require intervention

OTHER OUTCOMES:
Adverse event reporting | 1 year
  reporting of any adverse events that afflict study participants

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Willicombe, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No